CLINICAL TRIAL: NCT04873102
Title: A Phase II Single Center Single Arm Pilot Study Administering Danazol for Treatment of Cytopenias in Patients With Cirrhosis
Brief Title: Danazol for Treatment of Cytopenias in Patients With Cirrhosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Casey O'Connell, MD, Principal Investigator, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20-00366
Record Dates: First submitted 2020-12-09; First posted 2021-05-05 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cirrhosis, Liver; Cytopenia
MeSH Terms: conditions — Liver Cirrhosis; Cytopenia | interventions — Danazol

STUDY DESIGN:
Intervention Model Description: This is a phase II pilot study designed to assess the safety and efficacy of danazol for treatment of cytopenias in patients with CPC A/B cirrhosis. Subjects with telomere mutations and/or shortened telomeres will be treated with danazol 600 mg per day by mouth for a duration of 24 months. The goal will be to treat a total of 10 patients with telomere gene mutations and/or shortened telomere lengths.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Danazol in Treatment of Cytopenias (Experimental): AGENT: Danazol 600mg, Oral, Daily for 24 months
  Interventions: Drug: Danazol Pill

INTERVENTIONS:
Drug: Danazol Pill — Danazol is a synthetic steroid derived from ethisterone, It suppresses the pituitary-ovarian axis by inhibiting the pituitary output of gonadotropins. The pituitary-suppressive action of danazol is reversible. Danazol has been approved in treating endometriosis, fibrocystic breast disease, hereditary angioedema, thrombocytopenic purpura, and other conditions. It is metabolized and eliminated by renal and fecal pathways. The mean half-life of danazol in healthy males is 9.7 hours. After 6 months of 200 mg three times a day dosing in endometriosis patients, the half-life of danazol was reported as 23.7 hours.
  Adverse reactions from danazol include androgen like effects (i.e. weight gain, acne, mild hirsutism, edema, hair loss, voice change) and menstrual disturbances. The use of danazol in pregnancy is contraindicated. Other side effects include elevations in liver-enzyme levels and lipid abnormalities.
  Other Names: Danocrine

SUMMARY:
This is a phase II pilot study designed to assess the safety and efficacy of danazol for treatment of cytopenias in patients with CPC A/B cirrhosis. Subjects with or without telomere mutations and/or shortened telomeres will be treated with danazol 600 mg per day by mouth for a duration of 24 months. The goal will be to treat a total of 10 patients.

DETAILED DESCRIPTION:
Most studies estimate that between 6 and 77% of all patients with cirrhosis have abnormal hematologic indices (AHI), including anemia, thrombocytopenia and leukopenia. In a homogenous population of patients with compensated Child-Pugh Class (CPC) A/B cirrhosis, as many as 84% have AHI.18,19 The presence of AHI contributes to increased morbidity and mortality in a large proportion of cirrhotic patients. For example, thrombocytopenia can be a limiting factor when considering invasive surgical procedures due to the increased risk for bleeding. Leukopenia increases the risk for infections and chronic anemia contributes to worse outcomes after hemorrhagic episodes.18 Thrombocytopenia and leukopenia have been shown to be associated with death, transplant, clinical decompensation and hepatocellular carcinoma (HCC).19

The pathogenesis of AHI in patients with cirrhosis is often multifactorial, with splenic sequestration, portal hypertension, bone marrow suppression, and changes in hematopoietic stimulating factors contributing to the etiology.18 The severity of cytopenias does not consistently correlate with the degree of cirrhosis and may not correct after liver transplant. Current therapies have variable efficacy in improving cytopenias and management focuses primarily on supportive care with transfusions and growth factors.

Telomeres are repetitive DNA sequences located at the natural ends of linear chromosomes. They function to cap and protect chromosome ends from being recognized as damaged or infected DNA.3 During cell division, the "end-replication problem" arises as telomeres continually shorten because DNA polymerase cannot fully replicate the 3' end of chromosomes. The telomerase complex counters telomere attrition by elongating the telomere DNA after each cell division. Germline genetic defects in telomere maintenance and repair can cause dyskeratosis congenita, bone marrow failure, liver cirrhosis, pulmonary fibrosis, as well as increased susceptibility to various cancers. 4-5, 24-25

As a major complication of liver disease, cirrhosis is the main risk factor for progressive liver failure and HCC. To better understand the pathogenesis of cirrhosis, the connection between telomere attrition and cirrhosis has been examined in preclinical studies. Rudolph et al. found that telomerase reverse transcriptase (TERT)-deficient mice displayed reduced liver regeneration after partial hepatectomy and increased hepatic fibrosis after carbon tetrachloride exposure. After restoration of telomerase activity, there was improved liver function and cirrhosis reduction.21 Similarly, studies in humans found significantly accelerated telomere shortening and more telomere mutations in livers with cirrhosis and chronic hepatitis compared to normal livers.15 Patients with dyskeratosis congenita, pulmonary fibrosis, aplastic anemia, and short telomeres also showed an increased frequency of liver fibrosis and cirrhosis.

In an analysis of the Surveillance, Epidemiology and End Results (SEER)-Medicare database from 1992 through 2009, the development of liver disease was compared between 82,938 men with prostate cancer who did and did not undergo androgen deprivation therapy (ADT).12 Exposure to ADT was significantly associated with an increased subsequent risk of non-alcoholic fatty liver disease (54%), cirrhosis (35%) and any liver disease 47%). These data support a relationship between androgens and liver health, the mechanism of which is likely multifactorial

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and able to provide informed consent
* ECOG 0-2
* Compensated Child-Pugh class A of any etiology with the exception of chronic hepatitis B with one or more of the following cytopenias

  1. Leukopenia defined as white blood cell count <2000/mm3 or absolute neutrophil count <1000/mm3 along with thrombocytopenia <150,000/mm3 measured on two separate occasions at least 3 months apart within 6 months of enrollment
  2. Thrombocytopenia defined as platelet count <50,000/mm3 along with white blood cell count <4000/mm3 measured on two separate occasions at least 3 months apart within 6 months of enrollment
* Compensated Child-Pugh class B cirrhosis of any etiology with the exception of chronic hepatitis B with one or more of the following cytopenias:

  1. Leukopenia defined as white blood cell count ≤ 3500/mm3 measured on two separate occasions at least 3 months apart within 6 months of enrollment 3. Thrombocytopenia defined as platelet count ≤ 100,000/mm3 measured on two separate occasions at least 3 months apart within 6 months of enrollment
* Enrolled patients must have one or more of the following:

  * Presence of a genetic variant (defined as a known mutation, variant likely to be pathogenic or variant of undetermined significance with likely deleterious effect on transcription or translation) in at least one of the following genes: TERT, TERC, RTEL1, DKC, NOP10, NHP2, TINF2, WRAP53
  * Shortened telomere length in peripheral blood mononuclear cells (defined as age-adjusted telomere length at or below the 5th percentile)
  * Of note, patient's found to have telomere mutations know to confer a gain of function will be excluded
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception
* Women of childbearing potential (WOCBP) must have a negative serum test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of treatment

Exclusion Criteria:

* Cirrhosis secondary to chronic hepatitis B or any history of hepatitis B
* Patients with telomere related mutations know to confer gain of function will be excluded
* Patients known to be infected with HIV
* History of any hormone sensitive malignancy, including breast cancer, prostate cancer, hepatocellular carcinoma or liver adenoma as well as any patient considered high risk for developing malignancy (i.e. history of familial cancers including a first degree relative)
* Patients who are actively receiving anti-cancer therapy
* Liver decompensation event within the last 6 months (i.e. variceal bleed, ascites requiring paracentesis, hepatic encephalopathy)
* Active thrombosis or history of unprovoked thromboembolic disease, including cardiovascular events. If a patient has received and completed adequate anticoagulation for a provoked thrombosis, they can be included in the study.
* Pregnant or planning to become pregnant
* Females patients who are breast feeding
* Any contraindication to danazol use
* Uncontrolled co-morbid condition which would make the administration of danazol unsafe, including decompensated heart failure or known EF less than 40%, unstable angina pectoris, uncontrolled cardiac arrhythmia, decompensated liver failure, renal failure defined as creatinine greater than >1.6 or psychiatric illness that would limit compliance with study requirements
* Alanine aminotransferase and/or aspartate aminotransferase >3x upper limit of normal
* Alkaline phosphatase >2.5 x upper limit of normal
* Total bilirubin or direct bilirubin >2.5 x upper limit of normal
* Patients with known alcohol or drug abuse within the last year
* Concomitant use of hormone stimulants or hormone blocking agents.
* Concomitant use of other bone marrow stimulating agents that may affect white blood cell and platelet counts (i.e. G-CSF, romiplostim, eltrombopag, corticosteroids). Short term use of growth factors per standard of care in preparation for procedure or for other medical indications is acceptable. Patients taking corticosteroids above 5 mg of prednisone or the equivalent who are on a stable dose for at least 8 weeks prior to enrollment can be included.
* Concomitant treatment with systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Hematologic Response | 2 years
  Defined as normalization of WBC to ≥ 4000/µL or doubling of WBC from baseline, AND/OR normalization of platelet count to ≥150,000/µL or doubling of platelet count from baseline, from study entry to three months.
Occurrence of grade 3+ adverse events | Up to 2 years
  Adverse events will be measured using CTCAE v5 .

SECONDARY OUTCOMES:
Change in blood cell counts | 2 years
  Complete blood cell counts will be measured every 3 months for a total of 24 months
Change in peripheral blood telomere lengths | 2 years
  Telomere length will be measured at baseline and 24 months. Rate of telomere attrition will be measured and compared to age and sex matched controls.
Change in liver fibrosis | 2 years
  Liver fibrosis will be measured using transient elastrography (fibroscan) at baseline and 24 months
Change in liver function - Albumin | Up to 2 years
  Albumin level will be measured by blood test every 3 months from baseline to 24 months
Transplant-free survival | 2 years
  defined as time from study entry until liver transplant. Patients who have not undergone transplant will be censored at the time of last contact.
Overall survival | 2 years
  defined as the time from study entry until death. Patients who are alive at last follow-up will be censored.
Occurrence of clinical decompensation events | 2 years
  Number of decompensation events (i.e. variceal hemorrhage, ascites requiring intervention, and hepatic encephalopathy) will be counted during the 24 month study period and incidence calculated

CONTACTS AND LOCATIONS:
Overall Officials: Casey O'Connell, MD, Principal Investigator — Keck Hospital of USC
Locations (1):
- Keck Hosital of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT04873102/Prot_SAP_000.pdf